CLINICAL TRIAL: NCT01716559
Title: Multicenter, Observational Study to Evaluate NeoRecormon Treatment in Anemic Patients Suffering From Non-myeloid Malignancy Receiving Chemotherapy
Brief Title: An Observational Study of NeoRecormon (Epoetin Beta) in Anemic Patients With Non-myeloid Malignancy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25362
Record Dates: First submitted 2012-10-11; First posted 2012-10-30 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational, prospective, multicenter study will evaluate the treatment response rate and the safety of NeoRecormon (epoetin beta) in anemic patients with non-myeloid malignancy. In addition to NeoRecormon, patients receive chemotherapy for their malignancy. Data will be collected for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Presence of solid-tumor or non-myeloid malignancy
* Patients receiving chemotherapy
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Patients require NeoRecormon

Exclusion Criteria:

* Hypersensitivity to the drug
* Uncontrolled hypertension
* Female patients if pregnant and/or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anemic patients with non-myeloid malignancy
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Hungary (3):
  - Budapest
  - Kaposvár
  - Szolnok

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational study. A total of 160 participants were enrolled across 8 study centers in Hungary from 03 August 2010 to 28 March 2012.
Groups:
- Epoetin Beta: Participants receiving 30,000 International units (IU) of Epoetin beta (NeoRecormon) subcutaneously by prefilled pen injection once a week for 16 weeks were observed.
Period: Overall Study
Arm/Group | Epoetin Beta
Started | 160
Completed | 49
Not Completed | 111
Not completed — Adverse Event | 11
Not completed — Death | 21
Not completed — Withdrawal by Subject | 4
Not completed — Other withdrawal reason | 75

BASELINE CHARACTERISTICS:
Population: The Total population included all participants who met the inclusion and exclusion criteria and received at least one dose of study medication.
Groups:
- Epoetin Beta: Participants receiving 30,000 International units (IU) of Epoetin beta subcutaneously by prefilled pen injection once a week for 16 weeks were observed.
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Increase of Greater Than or Equal to 1 Gram Per Decilitre in Hemoglobin Level at Week 8
Description: Therapeutic response was defined as an increase of greater than or equal to (>=) 1 gram per decilitre (g/dL) in hemoglobin (Hb) level as compared to baseline, following 8 weeks of Epoetin beta treatment. The Therapeutic response rate was summarized as percentage of participants with an increase of >= 1 g/dL in Hb level at Week 8 as compared to baseline.
Time Frame: Baseline to Week 8
Population: The analysis was performed on total population. At the end of the Week 8, data allowing the evaluation of the therapeutic response was available for 103 participants out of total population of 160.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 103
percentage of participants | 67.96 [58.95 to 76.97]

2. Secondary Outcome: Mean Change From Baseline in Hemoglobin Level up to Week 16
Description: The mean change in Hb concentration was calculated by subtracting the baseline Hb concentration from the Weekly Hb concentration.
Time Frame: Baseline, Week 4, Week 8, Week 12, and Week 16
Population: The analysis was performed on Total population. The "n" signifies the number of participants assessed for mean change in hemoglobin level for specified time point.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 160
g/dL
  Week 4; n = 149 | 1.194 (0.133)
  Week 8, n = 103 | 1.641 (0.169)
  Week 12, n = 70 | 1.970 (0.198)
  Week 16, n = 50 | 1.789 (0.227)

3. Secondary Outcome: Percentage of Red Blood Cell Transfusion-free Participants
Description: Percentage of participants who have not received red blood cell (RBC) transfusion (packed RBC or whole blood) during the study were reported.
Time Frame: Up to Week 16
Population: The analysis was performed on Total population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 160
percentage of participants | 76.25 [69.66 to 82.84]

4. Secondary Outcome: Number of Participants With or With no Response on Efficacy of Treatment With or Without Iron Replacement Therapy
Description: Effect of individual iron supplementation on the efficacy of Epoetin beta treatment was described by percentage of participants with or with no response on efficacy of treatment due iron replacement therapy. Response was determined by calculating the difference in Hb level at H3 (Week 8) as compared to H1 (baseline). If H3-H1 is greater than (>) 1, there is a response (response value =1), otherwise there was no response (response value=0). If both were missing, then response was also missing. Response value as "1" denotes an effect on the response of treatment with or without iron replacement therapy. Response value as "0" denotes no effect on the response of treatment with or without iron replacement therapy.
Time Frame: Up to Week 16
Population: The analysis was performed on total population. At the end of the study, data allowing the evaluation of effect of individual iron supplementation on the efficacy of Epoetin beta treatment were available for 103 participants out of total population of 160.
Measure: Number; unit: participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 103
participants
  With IRT, Response value = 0 | 19
  With IRT, Response value = 1 | 44
  Without IRT, Response value = 0 | 9
  Without IRT, Response value = 1 | 31

5. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Number of participants with at least one AE and SAE were reported.
Time Frame: Up to Week 16
Population: The analysis was performed on total population.
Measure: Number; unit: participants
Arm/Group | Epoetin Beta
Number analyzed (Participants) | 160
participants
  Any AE | 43
  Any SAE | 25

ADVERSE EVENTS:
Time Frame: Up to Week 16
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Arm/Group | Epoetin Beta
Serious Adverse Events (participants affected / at risk) | 25/160
Other Adverse Events (participants affected / at risk) | 11/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Beta (N=160)
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Granulocytopenia (Blood and lymphatic system disorders) | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Disease progression (General disorders) | 9
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Brain abscess (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemiparesis (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Beta (N=160)
Anaemia (Blood and lymphatic system disorders) | 2
Granulocytopenia (Blood and lymphatic system disorders) | 3
Granulocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Metastasis to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights